CLINICAL TRIAL: NCT01272011
Title: Intermittent Hypoxia and Locomotor Training: Effects Following SCI
Brief Title: Effects of Breathing and Walking Treatments on Recovery Post-Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Florida (Other); Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B7182-W
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injuries; Brown Sequard; Central Cord Syndrome
Keywords: Respiration; Spinal cord injuries; Walking recovery
MeSH Terms: conditions — Spinal Cord Injuries; Central Cord Syndrome; Respiratory Aspiration | interventions — Respiratory Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1 Arm (Pilot) (Experimental): Individuals were exposed to intermittent hypoxia and locomotor training to establish our interventions (set up lab, train personnel, develop study protocols/interventions, etc)
  Interventions: Other: Intermittent Hypoxia; Other: Locomotor Training
- Phase 2 Arm (LTF) (Experimental): Individuals were exposed to 10 days of intermittent hypoxia to determine the effect of this intervention on ventilatory long-term facilitation, as measured by minute ventilation
  Interventions: Other: Intermittent Hypoxia
- Phase 3 Arm (Ventilatory Loading) (Other): Individuals were exposed to 10 days of intermittent hypoxia to determine changes in ventilatory loading.
  Interventions: Other: Intermittent Hypoxia

INTERVENTIONS:
Other: Intermittent Hypoxia — Individuals received exposure to intermittent hypoxia for 10 days, and placebo for 1-2 days.
  Other Names: Breathing Treatment
Other: Locomotor Training — Individuals received 10 days of locomotor training, intense walking training on a treadmill with body weight support. Manual assistance was provided at the legs to optimize stepping patterns.
  Arms: Phase 1 Arm (Pilot)

SUMMARY:
Change to Reflect What Was Done and reason Changes Were Made.

The purpose of this study is to determine (1) if a specific breathing treatment (intermittent hypoxia) can promote changes in breathing function and (2) if pairing breathing treatments (hypoxia) with locomotor training can enhance the benefits of walking recovery observed with locomotor training alone (without breathing treatments).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a very disabling health problem. Paralysis and paresis of limb and trunk muscles are major consequences of SCI and result in the inability to walk or difficulty walking. The most commonly stated goal by individuals with SCI during rehabilitation is the desire to walk again. Locomotor training (LT) that uses a body-weight support system and treadmill (BWST) is a task-specific rehabilitation intervention that allows practice of walking at normal speeds while loading the lower extremities, facilitating upright posture, and hip extension. Substantial improvement in ambulation can occur following locomotor training (LT) in individuals with motor incomplete spinal cord injury (iSCI). Despite these advances in activity-dependent rehabilitation, a need exists for defining complementary strategies that further amplify endogenous neuroplasticity. The proposed study will assess the therapeutic potential of (1) a respiratory training intervention (acute intermittent hypoxia, or AIH) on breathing function and (2) a combined locomotor (LT) and respiratory (AIH) training intervention for enhancing walking recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* At least 12 months post-incomplete spinal cord injury (I-SCI), including but not limited to the following syndromes: Brown Sequard and Central Cord Syndromes
* Upper motor neuron lesion (with upper motor neuron signs (i.e. presence of clonus, spasms, and/or hyperreflexia))
* A diagnosis of first time SCI including etiology from trauma, vascular, or orthopedic pathology
* Resting oxygen saturation (SpO2) levels of 95-99%
* Individuals who ambulate independently, with an assistive device, or who can walk when provided manual assistance
* Persons using anti-spasticity medication must maintain stable medication dosage during the study
* Able to give informed consent.
* Medical approval by individual's physician

Exclusion Criteria:

* Current participation in a rehabilitation program/research protocol that could interfere or influence the outcome measures of the current study
* History of congenital SCI (e.g. myelomeningocele, intraspinal neoplasm, Frederich's ataxia) or other degenerative spinal disorders (e.g. spinocerebellar degeneration, syringomyelia) that may complicate the protocol
* Inappropriate or unsafe fit of the harness due to the participant's body size and/or joint contractures or severe spasticity that would prohibit the safe provision of either training modality.
* Severe spasticity that would prohibit the safe provision of training.
* Pregnancy - all women of childbearing age will be required to undergo pregnancy testing prior to enrollment
* Unstable medical condition that could interfere with safety during participation in study (i.e. symptomatic cardiopulmonary complication, osteoporosis, contractures or other significant medical complications that would prohibit or interfere with testing of walking function and training or alter compliance with a training protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole J Tester, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

REFERENCES:
- [Derived] Tester NJ, Fuller DD, Fromm JS, Spiess MR, Behrman AL, Mateika JH. Long-term facilitation of ventilation in humans with chronic spinal cord injury. Am J Respir Crit Care Med. 2014 Jan 1;189(1):57-65. doi: 10.1164/rccm.201305-0848OC. PMID 24224903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from October, 2010 through April, 2014 through the North Florida/South Georgia VA Medical Center's Brain Rehabilitation Research Center.
Pre-assignment Details: Different study arms were carried out in different phases. The time individuals were enrolled determined which arm they were involved with. Participants enrolling knew which arm we currently were recruiting for. Individuals enrolled in early arms were invited back to other arms of the study if they chose--however, this was not a requirement.
Groups:
- Phase 1 Arm (Pilot): This group of participants were exposed to intermittent hypoxia and/or locomotor training. They were enrolled only to establish and streamline the protocol and train the laboratory personnel.
- Phase 2 Arm (LTF): This group of subjects were exposed to intermittent hypoxia and minute ventilation was recorded to determine whether ventilatory long term facilitation (LTF) was present.
- Phase 3 Arm (Ventilatory Loading): This group of subjects was exposed to intermittent hypoxia and ventilatory loading was assessed.
Period: Overall Study
Arm/Group | Phase 1 Arm (Pilot) | Phase 2 Arm (LTF) | Phase 3 Arm (Ventilatory Loading)
Started | 3 | 10 | 3
Completed | 3 | 8 | 3
Not Completed | 0 | 2 | 0
Not completed — Withdrawal By Subject or Failed Screen | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 Arm (Long Term Facilitation): This group of subjects were exposed to intermittent hypoxia and minute ventilation was recorded to determine whether ventilatory long term facilitation (LTF) was present.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Arm (Pilot) | Phase 2 Arm (Long Term Facilitation) | Phase 3 Arm (Ventilatory Loading) | Total
Number analyzed (Participants) | 3 | 8 | 3 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 2 | 11
  >=65 years | 0 | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 52 [52 to 52] | 53.13 [32 to 72] | 48.33 [26 to 67] | 51.86 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 0 | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 8 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Minute Ventilation - Phase 2
Description: Minute ventilation (Ve) is the volume of gas inhaled or exhaled from a person's lungs per minute. Minute ventilation during the end-recovery (ER) period at initial (i.e., Days 1 and 2, initial ER period) and final (i.e., Days 9 and 10, final ER period) days of the IH protocol were normalized to values from baseline with elevated carbon dioxide (B2) within each individual session to characterize daily effects of exposure to IH at the beginning and end of treatment. Values from baseline with elevated carbon dioxide and the ER period during the final days of the protocol (final B2 and final ER period, respectively) also were normalized to elevated carbon dioxide baseline during initial days of the protocol (initial B2) to describe the cumulative effects of repeated exposure to IH. Outcomes are reported as % increases in minute ventilation during initial and final treatment sessions for daily/acute effects and cumulative/chronic effects.
Time Frame: Pre- versus Post-treatment
Measure: Mean (Standard Error); unit: percentage of baseline
Arm/Group | Phase 1 Arm (Pilot) | Phase 2 Arm (LTF) | Phase 3 Arm (Ventilatory Loading)
Number analyzed (Participants) | 0 | 8 | 0
percentage of baseline
  Daily Acute Effects - Initial |  | 22.0 (5.2) |
  Daily Acute Effects - Final |  | 18.6 (3.6) |
  Cumulative Effects - Initial |  | 22.0 (5.2) |
  Cumulative Effects - Final |  | 22.1 (6.9) |
Statistical Analysis 1: Comparison: Phase 2 Arm (LTF); Daily acute and cumulative Pre vs Post comparisons; Test type: Superiority or Other; p < 0.001, Two-way RMANOVA Student-Newman-Keuls

2. Secondary Outcome: Ventilatory Loading - Phase 3
Description: Ventilatory load compensation was assessed in two ways. Mean slopes for (1) pressure vs. resistance (P vs R) and (2) airflow vs. resistance (AF vs R) were calculated for pre- and post-IH treatment.
Time Frame: Pre- versus Post-treatment
Population: Data were collected from 3 participants. However, clinical observations revealed results of interest from only 1/3 of the participants. Therefore, data from only this 1 individual were analyzed for presentation as a case study. The data from the other 2 participants were not analyzed.
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Phase 1 Arm (Pilot) | Phase 2 Arm (LTF) | Phase 3 Arm (Ventilatory Loading)
Number analyzed (Participants) | 0 | 0 | 1
unitless
  P vs R Baseline |  |  | -0.12 (0.02)
  P vs R Post Day 10 IH |  |  | -0.17 (0.02)
  AF vs R Baseline |  |  | -0.003 (0.001)
  AF vs R Post Day 10 IH |  |  | -0.0004 (0.002)
Statistical Analysis 1: Comparison: Phase 3 Arm (Ventilatory Loading); Compared outcomes from Baseline versus Post-Day 10 IH for mean slope of AF vs. Resistance; Test type: Superiority or Other; p < 0.05, RMANOVA and Student-Neuman-Keuls
Statistical Analysis 2: Comparison: Phase 3 Arm (Ventilatory Loading); Compared outcomes from Baseline versus Post-Day 10 IH for mean slope of of Pressure vs. Resistance; Test type: Superiority or Other; p < 0.05, RMANOVA and Student-Neuman-Keuls

ADVERSE EVENTS:
Arm/Group | Phase 1 Arm (Pilot) | Phase 2 Arm (Long Term Facilitation) | Phase 3 Arm (Ventilatory Loading)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/10 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes